CLINICAL TRIAL: NCT06401369
Title: CBCT-based Assessment of Apical Root Resorption and Alveolar Bone Height Following Orthodontic Treatment of Moderate Crowding With Labial vs. Lingual Fixed Appliances: A Randomized Controlled Trial
Brief Title: Comparing Labial and Lingual Orthodontic Appliances on Root Resorption and Bone Height
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-1-2024
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Crowding of Anterior Maxillary Teeth; Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The lingual fixed orthodontic group (LA) (Experimental): This group received treatment with lingual brackets with 0.018-inch slots (DTC Orthodontics, Hangzhou, China) applied with the aid of a special, indirect bonding technique, the "Modified HIRO® Technique." Individual lingual archwires (Forestadent®, Germany) were also used.
  Interventions: Procedure: Lingual brackets
- The labial fixed orthodontic group (BA) (Active Comparator): Patients in this group received treatment with labial appliances with 0.018-inch slots (American Orthodontics brackets, Mini Master series, MBT prescription) directly bonded on both arches. Prefabricated archwires (American Orthodontics, Sheboygan, WI, USA) were also used.
  Interventions: Procedure: Buccal brackets

INTERVENTIONS:
Procedure: Lingual brackets — These brackets will be used on the lingual surfaces of the upper and lower teeth.
  Arms: The lingual fixed orthodontic group (LA)
Procedure: Buccal brackets — These brackets will be used on the vestibular surfaces of the upper and lower teeth.
  Arms: The labial fixed orthodontic group (BA)

SUMMARY:
Patients who have moderate crowding that could be treated on a non-extraction will be treated in this study. The apical root resorption and alveolar bone height of the lingual and labial fixed appliances will be assessed. All patients will receive a cone-beam computed tomography (CBCT) scan at two different times (T0: Before treatment, T1: After treatment).

There are two groups: The first group (Experimental): The patients in this group will be treated using Lingual Fixed Orthodontic Appliances. The second group (Control): The patients in this group will be treated using Labial Fixed Orthodontic Appliances.

DETAILED DESCRIPTION:
Recently, the therapeutic results of lingual orthodontics have become similar to those produced by labial orthodontics. However, lingual appliances act differently. The application of force near the center of resistance and the distance between the lingual brackets leads to an increase in friction and, thus, an increase in the force applied during treatment. In addition, the contact of the lower incisors with the brackets of the upper incisors in the lingual technique can lead to the intrusion of these incisors. Therefore, these factors can be potential risks for apical root resorption and alveolar bone height in lingual orthodontics.

2D radiographs may not accurately depict the true amount of root resorption due to magnification errors and difficulties in obtaining repeatable images. Besides, conventional two-dimensional radiographs cannot accurately assess alveolar bone height in the anterior region. CBCT has proven to be valuable in diagnosing root resorption due to its capability to produce distortion-free images, as well as its ability to maintain a high level of reproducibility despite changes in tooth positions after treatment, with high sensitivity and specificity. On the other hand, the use of CBCT allows for an evaluation of alveolar bone height in the anterior region with high accuracy and precision.

ELIGIBILITY:
Inclusion Criteria:

1. Class I molar and canine relationships on both sides.
2. Moderate crowding of both arches of about 4 to 6 mm treated on a non-extraction basis.
3. Age from 18 to 25 years.
4. The presence of permanent dentition (except third molars).

Exclusion Criteria:

1. The existence of craniofacial syndromes, cleft lip and/or palate (soft and/or hard).
2. Skeletal or dental crossbite.
3. Patients with missing teeth or periodontal diseases.
4. Previous orthodontic treatment.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in tooth lengths | T0: one day before the commencement of treatment. T1: one day following the end of treatment
  Axial, coronal, and sagittal planes of the CBCT images will be reoriented to be perpendicular to the long axis of each tooth under assessment. The distances were measured as follows.
  Central and lateral incisors: from incisal edge to apex (sagittal section). Canines: from cusp tip to apex (sagittal section). Single-rooted premolar: from vestibular cusp tip to apex (sagittal section). Two-rooted premolar: from vestibular cusp tip to apex (sagittal section) and lingual cusp tip to apex (coronal section).
  Upper molars: from the mesiolingual cusp tip to the apex of the lingual root of the molar (coronal section), from the mesobuccal cusp tip to the apex of the mesobuccal root of the molar (sagittal section), from distobuccal cusp tip to the apex of distobuccal root of molar (sagittal section).
Change in the alveolar bone height | T0: one day before the commencement of treatment. T1: one day following the end of treatment
  The CBCT images were redirected according to the long axis of each tooth as given previously.
  The distance between the cementoenamel junction and the crest of the alveolar bone was measured in the sagittal plane for central and lateral incisors, while in the coronal plane for canines. For the premolars and first molars, the distance between the cementoenamel junction and the crest of the alveolar bone was measured in the coronal plane.

CONTACTS AND LOCATIONS:
Overall Officials: Jehad M. Kara-Boulad, DDS MSc PhD, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Ahmad S. Burhan, DDS MSc PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khattab TZ, Farah H, Al-Sabbagh R, Hajeer MY, Haj-Hamed Y. Speech performance and oral impairments with lingual and labial orthodontic appliances in the first stage of fixed treatment. Angle Orthod. 2013 May;83(3):519-26. doi: 10.2319/073112-619.1. Epub 2012 Oct 18. PMID 23075062
- [Background] Kara-Boulad JM, Burhan AS, Hajeer MY, Khattab TZ, Nawaya FR. Evaluation of the Oral Health-Related Quality of Life (OHRQoL) in Patients Undergoing Lingual Versus Labial Fixed Orthodontic Appliances: A Randomized Controlled Clinical Trial. Cureus. 2022 Mar 22;14(3):e23379. doi: 10.7759/cureus.23379. eCollection 2022 Mar. PMID 35371870
- [Background] Nassif CE, Cotrim-Ferreira A, Conti ACCF, Valarelli DP, de Almeida Cardoso M, de Almeida-Pedrin RR. Comparative study of root resorption of maxillary incisors in patients treated with lingual and buccal orthodontics. Angle Orthod. 2017 Nov;87(6):795-800. doi: 10.2319/041117-247.1. Epub 2017 Jul 24. PMID 28737425
- [Background] Hajeer MY, Al-Homsi HK, Alfailany DT, Murad RMT. Evaluation of the diagnostic accuracy of CBCT-based interpretations of maxillary impacted canines compared to those of conventional radiography: An in vitro study. Int Orthod. 2022 Jun;20(2):100639. doi: 10.1016/j.ortho.2022.100639. Epub 2022 May 21. PMID 35606269
- [Background] Alfailany DT, Shaweesh AI, Hajeer MY, Brad B, Alhaffar JB. The diagnostic accuracy of cone-beam computed tomography and two-dimensional imaging methods in the 3D localization and assessment of maxillary impacted canines compared to the gold standard in-vivo readings: A cross-sectional study. Int Orthod. 2023 Sep;21(3):100780. doi: 10.1016/j.ortho.2023.100780. Epub 2023 Jun 6. PMID 37290351
- [Background] Kara-Boulad JM, Burhan AS, Hajeer MY, Khattab TZ, Nawaya FR, Al-Sabbagh R. Treatment of Moderately Crowded Teeth Using Lingual Fixed Appliance Prepared by a Modified HIRO(R) Technique: A Case Report and Method Description. Cureus. 2022 May 17;14(5):e25077. doi: 10.7759/cureus.25077. eCollection 2022 May. PMID 35600066